CLINICAL TRIAL: NCT02005276
Title: A Randomized Trial of Behavioral Economic Interventions to Improve Physical Activities: Lottery Incentives
Brief Title: Way to Be Active 2 (Lotteries)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 819103
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Sedentary Employees
Keywords: Sedentary; Behavioral Economic Intervention; Team Studies; Financial Incentives; Workplace Wellness; Team Incentives
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (No Intervention): Participants receive either an email or text message daily (based on the participant's preference) stating whether the participant achieved the 7000 step goal during the previous day.
- Basic Lottery (Experimental): Participants receive either an email or text message daily (based on the participant's preference) stating whether the participant achieved the 7000 step goal during the previous day. Each day a lottery will be held, and participants will be eligible to collect monetary rewards only if the participant met the step goal the day before. The names of the winners will be announced during each lottery. The daily lotteries are as follows:
  About a 1 in 4 chance of winning $5. Expected value is about $1.40 per person per day.
  Interventions: Behavioral: Basic Lottery
- Combined Lottery (Experimental): Participants receive either an email or text message daily (based on the participant's preference) stating whether the participant achieved the 7000 step goal during the previous day. Each day a lottery will be held, and participants will be eligible to collect monetary rewards only if the participant met the step goal the day before. The names of the winners will be announced during each lottery. The daily lotteries are as follows:
  About a 1 in 5 chance of winning $5 and a 1 in 100 chance of winning $50. Expected value is about $1.40 per person per day.
  Interventions: Behavioral: Combined Lottery
- Jackpot Lottery (Experimental): Participants receive either an email or text message daily (based on the participant's preference) stating whether the participant achieved the 7000 step goal during the previous day. Each day a lottery will be held, and participants will be eligible to collect monetary rewards only if the participant met the step goal the day before. The names of the winners will be announced during each lottery. The daily lotteries are as follows:
  About a 1 in 400 chance of winning $500. Expected value is about $1.40 per person per day.
  Interventions: Behavioral: Jackpot Lottery

INTERVENTIONS:
Behavioral: Basic Lottery — Participants who meet their daily step goals will be eligible for a daily lottery. They will have about a 1 in 4 chance of winning $5. Expected value is about $1.40 per person per day.
  Arms: Basic Lottery
Behavioral: Combined Lottery — Participants who meet their daily step goals will be eligible for a daily lottery. They will have about a 1 in 4 chance of winning $5 and a 1 in 100 chance of winning $50. Expected value is about $1.40 per person per day.
  Arms: Combined Lottery
Behavioral: Jackpot Lottery — Participants who meet their daily step goals will be eligible for a daily lottery. They will have about a 1 in 400 chance of winning $500. Expected value is about $1.40 per person per day.
  Arms: Jackpot Lottery

SUMMARY:
Employers are increasingly looking for opportunities to motivate sedentary employees to become more physically active. Workplace walking programs have had mixed success and typically show most improvement among participants that are already fairly active at a baseline. The goal of this study is to determine whether a financial incentive program can motivate sedentary employees to increase the number of steps they walk per day to meet a minimum threshold.

Our primary outcome measure is the proportion of days a minimum activity of 7000 steps or more is achieved. We will assess outcomes each week for 3 months using incentives followed by 3 months of follow-up without incentives. Secondary outcomes will include the average steps walked per day.

ELIGIBILITY:
Inclusion Criteria:

* 1. We will use a minimum age of 18 to ensure all individuals are legally able to consent.
* 2. Participant will need an iPhone or Android smartphone to be able to use the Moves App for tracking steps

Exclusion Criteria:

* Conditions that would make participation infeasible: 1a. Inability to consent 1b. Illiteracy and/or inability to speak, read, and write English 1c. Participation in another research study 2. Conditions that would make participation unsafe: 2a. Current treatment for drug or alcohol use 2b. Consumption of at least 5 alcoholic drinks per day 2c. Myocardial infarction or stroke within the past 6 months 2d. Current addiction to prescription medicines or street drugs 2e. Serious psychiatric diagnoses (e.g., severe major depressive disorder, bipolar disorder, schizophrenia) 2f. Pregnant or currently breastfeeding 2g. Metastatic cancer 2h. Unstable medical conditions that would likely prevent the participant from completing the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2014-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Volpp, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Basic Lottery: Participants receive either an email or text message daily (based on the participant's preference) stating whether the participant achieved the 7000 step goal during the previous day. Each day a lottery will be held, and participants will be eligible to collect monetary rewards only if the participant met the step goal the day before. The names of the winners will be announced during each lottery. The daily lotteries are as follows:
  About a 1 in 4 chance of winning $5. Expected value is about $1.40 per person per day.
  Basic Lottery: Participants who meet their daily step goals will be eligible for a daily lottery. They will have about a 1 in 4 chance of winning $5. Expected value is about $1.40 per person per day.
- Jackpot Lottery: Participants receive either an email or text message daily (based on the participant's preference) stating whether the participant achieved the 7000 step goal during the previous day. Each day a lottery will be held, and participants will be eligible to collect monetary rewards only if the participant met the step goal the day before. The names of the winners will be announced during each lottery. The daily lotteries are as follows:
  About a 1 in 400 chance of winning $500. Expected value is about $1.40 per person per day.
  Jackpot Lottery: Participants who meet their daily step goals will be eligible for a daily lottery. They will have about a 1 in 400 chance of winning $500. Expected value is about $1.40 per person per day.
- Combined Lottery: Participants receive either an email or text message daily (based on the participant's preference) stating whether the participant achieved the 7000 step goal during the previous day. Each day a lottery will be held, and participants will be eligible to collect monetary rewards only if the participant met the step goal the day before. The names of the winners will be announced during each lottery. The daily lotteries are as follows:
  About a 1 in 5 chance of winning $5 and a 1 in 100 chance of winning $50. Expected value is about $1.40 per person per day.
  Combined Lottery: Participants who meet their daily step goals will be eligible for a daily lottery. They will have about a 1 in 4 chance of winning $5 and a 1 in 100 chance of winning $50. Expected value is about $1.40 per person per day.
Period: Overall Study
Arm/Group | Control | Basic Lottery | Jackpot Lottery | Combined Lottery
Started | 65 | 41 | 59 | 44
Completed Intervention | 61 | 39 | 56 | 42
Completed (Completed follow-up) | 60 | 39 | 56 | 41
Not Completed | 5 | 2 | 3 | 3
Not completed — No longer interested | 5 | 2 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Basic Lottery | Jackpot Lottery | Combined Lottery | Total
Number analyzed (Participants) | 65 | 41 | 59 | 44 | 209
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (11.0) | 41.2 (11.1) | 40.6 (10.5) | 42.9 (10.3) | 41.2 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 32 | 44 | 33 | 161
  Male | 13 | 9 | 15 | 11 | 48
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 33.8 (6.0) | 32.0 (4.8) | 33.5 (4.9) | 32.9 (4.3) | 33.2 (5.0)
Race/ethnicity [Count of Participants; unit: Participants]
  White non-Hispanic | 45 | 30 | 36 | 34 | 145
  African American non-Hispanic | 12 | 7 | 12 | 8 | 39
  Other non-Hispanic | 5 | 2 | 5 | 2 | 14
  Hispanic | 3 | 2 | 6 | 0 | 11
Education [Count of Participants; unit: Participants]
  Less than college | 1 | 1 | 4 | 4 | 10
  Some college | 13 | 9 | 11 | 11 | 44
  College graduate | 51 | 31 | 44 | 29 | 155
Marital status [Count of Participants; unit: Participants]
  Single | 23 | 14 | 14 | 17 | 68
  Married | 32 | 16 | 37 | 22 | 107
  Other | 10 | 11 | 8 | 5 | 34
Annual household income [Count of Participants; unit: Participants]
  Less than $50,000 | 17 | 12 | 12 | 8 | 49
  $50,000 to $100,000 | 22 | 18 | 22 | 25 | 87
  Greater than $100,000 | 21 | 9 | 19 | 8 | 57
  Missing | 5 | 2 | 6 | 3 | 16
Iphone smartphone [Count of Participants; unit: Participants] | 43 | 30 | 38 | 27 | 138

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Days a Minimum Activity of 7000 Steps or More is Achieved During Intervention
Description: Our primary outcome measure is the proportion of days a minimum activity of 7000 steps or more is achieved. We will assess outcomes for 3 months using incentives followed by 3 months of follow-up without incentives. All available data will be analyzed, and missing will be treated as true missing data points. Secondary outcomes will include the average steps walked per day.
Time Frame: End of study- 6 months of after enrollment
Measure: Mean (95% Confidence Interval); unit: Proportion of participant days
Arm/Group | Control | Basic Lottery | Jackpot Lottery | Combined Lottery
Number analyzed (Participants) | 65 | 41 | 59 | 44
Proportion of participant days
  Intervention Period (3 months with incentives) | 0.264 [0.192 to 0.336] | 0.319 [0.227 to 0.410] | 0.290 [0.216 to 0.365] | 0.384 [0.298 to 0.470]
  Follow Up Period (3 months without incentives) | 0.191 [0.134 to 0.249] | 0.211 [0.138 to 0.284] | 0.155 [0.096 to 0.215] | 0.215 [0.144 to 0.286]

2. Secondary Outcome: Average Number of Steps Per Day During Intervention
Description: Secondary outcomes include average number of steps per day during intervention (with incentives) and follow up periods (without incentives).
Time Frame: End of study- 6 months after enrollment
Measure: Mean (95% Confidence Interval); unit: steps per day
Arm/Group | Control | Basic Lottery | Combined Lottery | Jackpot Lottery
Number analyzed (Participants) | 65 | 41 | 44 | 59
steps per day
  Intervention Period (3 months with incentives) | 4744.8 [4128.7 to 5360.9] | 5022.9 [4238.4 to 5807.4] | 5439.6 [4703.2 to 6175.9] | 4838.0 [4200.3 to 5475.7]
  Follow Up Period (3 months without incentives) | 4068.9 [3486.7 to 4651.1] | 4408.4 [3669.4 to 5147.4] | 4449.5 [3730.2 to 5168.8] | 3800.3 [3197.4 to 4404.2]

ADVERSE EVENTS:
Arm/Group | Control | Basic Lottery | Jackpot Lottery | Combined Lottery
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/41 | 0/59 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/41 | 0/59 | 0/44
Other Adverse Events (participants affected / at risk) | 0/65 | 0/41 | 0/59 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No